CLINICAL TRIAL: NCT03286335
Title: Local Control, Quality of Life and Toxicities in Adults With Benign or Indolent Brain Tumors Undergoing Proton Radiation Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Helen A. Shih, MD, Shih, Helen A, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-250
Record Dates: First submitted 2017-09-12; First posted 2017-09-18 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Brain Tumor
Keywords: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Proton Radiation (Experimental): * Radiation therapy will be delivered typically five (5) days per week on weekdays
  * Proton Radiation dose be determine by histology
  Interventions: Radiation: Proton Radiation

INTERVENTIONS:
Radiation: Proton Radiation — Radiation treatment

SUMMARY:
This research study is studying Proton Radiation as a possible treatment for brain tumor.

The radiation involved in this study is:

-Proton Radiation

DETAILED DESCRIPTION:
The main purpose of this study is to see how well the tumor is responding to the Proton Radiation up to 5 years after the participant receive it. The investigators are also looking for how this type of radiation affects the quality of life as well as any type of side effect the participant may have after the radiation is administered.

The FDA (the U.S. Food and Drug Administration) has not approved Proton Radiation for this specific disease but it has been approved for other uses.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven benign or malignant brain tumor requiring tumor bed or tumor irradiation. This may include, but is not limited to, low-grade or favorable high-grade glioma, pituitary adenoma, vestibular schwannoma (acoustic neuroma), and meningioma as the most common diagnoses. Other tumor types that require irradiation and are deemed appropriate for proton radiation therapy are also eligible. Patients with a presumed diagnosis based on imaging and clinical characteristics will be permitted on this trial without pathological diagnostic confirmation if it is within standard of care to offer radiation therapy without a biopsy.
* Participants must otherwise be indicated for proton radiation therapy
* Age 18 years or older
* Karnofsky performance status ≥ 60 (see Appendix A)
* Participants may have had any extent of prior surgery and/or chemotherapy.
* Must be able to speak and comprehend English
* Ability to understand and willingness to sign a written informed consent document
* The effects of proton radiation therapy on the developing human fetus are known to be teratogenic. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study treatment, and 4 months after completion of proton therapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study treatment, and 4 months after completion of proton therapy.
* Life expectancy greater than or equal to 6 months.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or lactating women are excluded from this study because radiation is known to have teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with radiation therapy, breastfeeding should be discontinued if the mother is treated with radiation therapy.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 3 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-26 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Duration of Local Control | 2 years
  The duration of local control will be measured from the start date of protocol radiation until the date of progressive disease. Local control is defined as the lack of tumor growth as determined by a brain MRI (magnetic resonance imaging). This will include tumors that appear unchanged in size as compared to the baseline pre-radiation scan and also tumors that appear slightly reduced in size as may occur in response to radiation therapy. Inflammation secondary to radiation therapy can radiographically mimic subtle disease progression and may need to be confirmed with serial imaging.
  Progression is defined as an increase in the size of the tumor, a significant increase in T2/FLAIR non-enhancing lesion on sable or increasing doses of corticosteroids compared to baseline, the appearance of any new lesion, clear clinical deterioration not attributable to any other cause apart from the tumor, or failure to return for evaluation due to death or deteriorating condition.

SECONDARY OUTCOMES:
Quality of Life Assessment EORTC-QLQ-C30 | 2 years
  Quality of life in relation to overall physical functioning will be assessed using the European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaires (QLQ). Overall functioning will be assessed at baseline and follow-up evaluations using EORTC-QLQ-C30.
  Mixed effects models will be used to analyze the repeated measures of EORTC-QLQ with participant-specific intercepts and slopes assumed as random effects. Tumor type will be modeled as fixed effects in order to estimate quality of life changes over time among participants with each benign and malignant diagnosis.
Quality of Life Assessment EORTC-QLQ-BN20 | 2 Years
  Quality of life in relation to symptoms specific to brain cancer will be assessed using the European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaires (QLQ). Brain cancer-specific symptoms will be assessed at baseline and follow-up evaluations using EORTC-QLQ-BN20.
  Mixed effects models will be used to analyze the repeated measures of EORTC-QLQ with participant-specific intercepts and slopes assumed as random effects. Tumor type will be modeled as fixed effects in order to estimate quality of life changes over time among participants with each benign and malignant diagnosis.
Quality of Life Assessment HADS | 2 Years
  State anxiety and depression will be measured with the Hospital Anxiety and Depression Scale (HADS). HADS screens for mood disorders in medically ill participants; it focuses on subjective rather than physical symptoms, which may be confounded with illness.
  Mixed effects models will be used to analyze the repeated measures of HADS with participant-specific intercepts and slopes assumed as random effects. Tumor type will be modeled as fixed effects in order to estimate mood changes over time among participants with each benign and malignant diagnosis.
Vision Loss | 2 years
  Those participants determined to have had proton radiation exposure to any part of the optic pathway that could potentially affect vision will undergo standard afferent neuro-ophthalmological evaluation, which includes tests of visual acuity, color perception, pupillary function, visual field testing, and optic disc appearance. Participants with any tumor type will be evaluable for visual outcome if the battery of neuro-ophthalmology evaluation were performed at baseline. Testing will be discontinued if the participant becomes blind.
  The cumulative incidence of developing vision loss among evaluable participants will be analyzed with failure defined as decline in one or more of the vision function tests and with competing risks of progressive disease and death.
Ototoxicity | 2 years
  For participants with proton radiation exposure to the skull base audiologic system, standard audiologic testing will be performed, unless poor hearing inadequate for useful function is present at baseline. Testing will be discontinued if the participant becomes deaf. Participants with any tumor type will be evaluable for hearing outcome if audiology evaluation were performed at baseline.
  The cumulative incidence of developing ototoxicity among evaluable participants will be analyzed with failure defined as significant decrease in Pure Tone Average or/and Word Recognition Score and with competing risks of progressive disease and death
Neuroendocrine dysfunction | 2 years
  Participants will be candidates for neuroendocrine testing if they were determined to have any radiation exposure to the hypothalamus or pituitary gland or to have a target lesion within 2 cm of either of these normal structures, unless panhypopituitarism is present at baseline. Participants with any tumor type will be evaluable for endocrine outcome if neuroendocrine evaluation were performed at baseline.
  The cumulative incidence of developing neuroendocrine dysfunction among evaluable participants will be analyzed with failure defined as any hormonal deficiency confirmed by test criteria and with competing risks of progressive disease and death.
Neurocognitive effects | 2 years
  Participants with any tumor type will be evaluable for neurocognitive analysis if the optional neuropsychological evaluation were performed at baseline and/or at least one follow-up. Mixed effects models will be used to analyze the repeated measures of intelligence, language, visuospatial/motor functioning, learning/memory and attention/executive functioning, with participant-specific intercepts and slopes assumed as random effects. Tumor and treatment characteristics may be modeled as fixed effects in order to estimate their effects on neurocognitive changes over time.
Alopecia | 2 years
  Participants with any tumor type will be evaluable for alopecia unless they are virtually bald at baseline and graded using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Maximal hair loss will be documented between the last week of radiation and 4 weeks later, while permanent hair loss will be defined at 2 years post-treatment.
CD4 count | 2 years
  Participants with any tumor type will be evaluable for CD4 analysis if they were to consent to the optional assessment of CD4 count. The worst grade of CD4 count will be defined using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 during the short term (on-treatment and 1 to 3 months post-radiation) and long term (6 months to 2 years post-radiation).

CONTACTS AND LOCATIONS:
Overall Officials: Helen A Shih, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No